CLINICAL TRIAL: NCT07402096
Title: Effect of a Mindfulness-Based Stress Reduction Program on Hot Flashes and Sleep Quality in Menopausal Women: A Randomized Controlled Trial
Acronym: MBSR-MENO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Kader ATABEY, Kader ATABEY, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INU-MBSR-MEN-2025
Record Dates: First submitted 2025-12-30; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Menopause; Hot Flashes; Sleep Wake Disorders
Keywords: Menopause; Hot Flashes; Non-pharmacological intervention
MeSH Terms: conditions — Hot Flashes; Sleep Wake Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (MBSR) Group (Experimental): Participants in this arm will receive an 8-week Mindfulness-Based Stress Reduction (MBSR) program. The program consists of weekly sessions lasting 60-90 minutes and includes mindfulness practices such as breathing awareness, body scan, emotional awareness, stress response awareness, and mindfulness in daily life. Sessions will be delivered through a combination of face-to-face and online formats.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Control Group (No Intervention): Participants in this arm will receive no intervention during the study period and will continue with their usual care. They will complete the same outcome assessments as the intervention group at baseline and at the end of the study.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Mindfulness-Based Stress Reduction (MBSR) is a structured behavioral intervention consisting of an 8-week program with weekly sessions lasting 60-90 minutes. The program includes mindfulness practices such as breathing awareness, body scan, emotional awareness, stress response awareness, and mindfulness in daily life. Sessions are delivered through a combination of face-to-face and online formats.
  Arms: Mindfulness-Based Stress Reduction (MBSR) Group

SUMMARY:
Menopause is a natural transition characterized by vasomotor symptoms such as hot flashes and sleep disturbances, which can significantly impair quality of life. Non-pharmacological interventions are increasingly recommended for women who cannot or prefer not to use hormone therapy. Mindfulness-Based Stress Reduction (MBSR) is a structured behavioral intervention that has shown beneficial effects on stress-related symptoms and sleep quality; however, evidence regarding its effects on menopausal symptoms remains limited.

This randomized controlled trial aims to evaluate the effectiveness of an 8-week MBSR program on hot flash frequency and severity and sleep quality in menopausal women. A total of 90 menopausal women will be randomly assigned to either an intervention group receiving the MBSR program or a control group receiving no intervention. Participants in the intervention group will attend weekly sessions and engage in mindfulness practices, including breathing awareness, body scan, and stress management techniques.

Primary outcomes include changes in hot flash frequency and severity and sleep quality, assessed using validated self-report measures. The findings of this study are expected to contribute to evidence-based, non-pharmacological management strategies for menopausal symptoms.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial with a pretest-posttest control group design to evaluate the effects of an 8-week Mindfulness-Based Stress Reduction (MBSR) program on menopausal symptoms. The study population consists of menopausal women aged 45-60 years who report experiencing hot flashes and poor sleep quality.

Participants will be recruited from gynecology outpatient clinics and randomly assigned to either the intervention group or the control group. The intervention group will participate in an 8-week standardized MBSR program consisting of weekly sessions lasting 60-90 minutes. The program includes mindfulness practices such as breathing awareness, body awareness, emotional regulation, stress response awareness, and mindfulness in daily life. Sessions will be delivered through a combination of face-to-face and online formats. The control group will not receive any intervention during the study period.

Outcome measures will be assessed at baseline and at the end of the 8-week intervention period. Primary outcome measures include hot flash frequency and severity and sleep quality, assessed using validated instruments. Secondary outcomes include mindfulness levels and perceived symptom-related distress. Data will be analyzed using appropriate statistical methods to compare within-group and between-group changes. Ethical approval has been obtained, and written informed consent will be obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* - Women aged between 45 and 60 years
* Postmenopausal status defined as at least 12 months since the last menstrual period
* Presence of hot flashes
* Poor sleep quality (Pittsburgh Sleep Quality Index score >5)
* Ability to understand and complete questionnaires
* Access to the internet and ability to use a smartphone or computer for online sessions
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Current use of hormone replacement therapy

  * Use of psychiatric medications
  * Diagnosis of a psychiatric disorder
  * Severe hearing or visual impairment
  * Previous participation in mindfulness-based or yoga programs
  * Incomplete baseline assessments
  * Failure to attend intervention sessions

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hot Flash Frequency and Severity | Baseline and 8 weeks
  Change from baseline to 8 weeks in hot flash frequency and severity, assessed using a validated hot flash diary or hot flash rating scale. Higher scores indicate greater symptom severity.
Change in Sleep Quality | Baseline and 8 weeks
  Change in sleep quality from baseline to 8 weeks, assessed using the Pittsburgh Sleep Quality Index (PSQI). Higher scores indicate poorer sleep quality.